CLINICAL TRIAL: NCT04283890
Title: Phase1b/2 Study Combining Hepatic Percutaneous Perfusion With Ipilimumab Plus Nivolumab in Advanced Uveal Melanoma
Brief Title: PHP and Immunotherapy in Metastasized UM
Acronym: CHOPIN
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, HW Kapiteijn, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NL69508.058.19
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Uveal Melanoma, Metastatic
Keywords: Advanced uveal melanoma; Percutaneous Hepatic Perfusion; Immunotherapy
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: In the phase 1b part, safety and feasibility of combining percutaneous hepatic perfusion with 4 courses of ipilimumab and nivolumab will be investigated. In the randomized phase 2 part, efficacy as measured by progression-free survival at one year comparing PHP only versus PHP plus ipilimumab/nivolumab will be evaluated.
Masking Description: Open label, single center, phase Ib/randomized phase II trial, evaluating the safety and efficacy (as measured by RECIST 1.1) of the combination of PHP and ipilimumab/nivolumab in patients with unresectable hepatic and extrahepatic metastases of uveal melanoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase Ib (Experimental)
  Interventions: Drug: Ipilimumab and nivolumab; Drug: Melphalan chemosaturation via percutaneous hepatic perfusion
- Phase II - Combination treatment (Active Comparator)
  Interventions: Drug: Ipilimumab and nivolumab; Drug: Melphalan chemosaturation via percutaneous hepatic perfusion
- Phase II - PHP (Active Comparator)
  Interventions: Drug: Melphalan chemosaturation via percutaneous hepatic perfusion

INTERVENTIONS:
Drug: Ipilimumab and nivolumab — The effect of ipilimumab and nivolumab has previously been tested in metastatic uveal melanoma. In this study the combination with percutaneous hepatic perfusion will be performed in order to evaluate the effect.
  Arms: Phase II - Combination treatment; Phase Ib
Drug: Melphalan chemosaturation via percutaneous hepatic perfusion — The effect of ipilimumab and nivolumab has previously been tested in metastatic uveal melanoma. In this study the combination with percutaneous hepatic perfusion will be performed in order to evaluate the effect.

SUMMARY:
Melanoma of the eye (ocular/uveal melanoma) is an uncommon type of cancer that is associated with a high mortality. It usually disseminates rapidly throughout the body, most commonly to the liver and lungs. In this study a combination therapy with immunotherapy (ipilimumab with nivolumab) and chemotherapy (melphalan) will be assessed for the treatment of disseminated uveal melanoma. Melphalan will be administered selectively to the liver via percutaneous hepatic perfusion, limiting the systemic effect of chemotherapy. With this treatment combination we aim to find a treatment for disseminated uveal melanoma, both in the liver as in the other organs.

DETAILED DESCRIPTION:
Uveal melanoma (UM) is an uncommon malignancy (0.6-0.7 cases/100.000/year) that, in the case of metastatic stage, has a poor prognosis for response to treatment and survival. It is remarkable for its purely hematogenous pattern of dissemination, most commonly to the liver (60%) and lungs (25%). Current approaches using percutaneous hepatic perfusion (PHP) with melphalan resulted in response rates of up to 40% in the liver (1, 2) (for results of our own phase II study see paragraph 6.3.2). However, a main part of the patients developed extrahepatic disease in the follow-up, whereas the liver metastases were mainly stable.

Checkpoint inhibitors have been shown to improve overall survival in metastasized cutaneous melanoma in phase III studies (3-6), but seem to have limited activity as monotherapies in metastasized uveal melanoma (7-9). The combination of ipilimumab and nivolumab has achieved 2 out of 6 patients PR in a retrospective analysis (10). Interestingly, both patients had a liver-directed therapy (SIRT and chemoembolization) before the immunotherapy.

Combination of radio-frequency ablation (RFA) and anti-CTLA-4 enhanced antigen-loading of dendritic cells, and induced long-lasting anti-tumor immune responses in a murine melanoma model without induction of any severe side effects (11, 12). A phase Ib/II trial by Blank et al. (13) showed unconfirmed responses in some patients when RFA was combined with ipilimumab in uveal melanoma, but long-term disease stabilization was not achieved. Most of the responses were seen in extrahepatic metastases. Combining percutaneous hepatic perfusion (PHP) with checkpoint inhibitors could together lead to control of hepatic and extrahepatic disease. Therefore, we propose the current trial: Phase1b/2 Study Combining Hepatic Percutaneous Perfusion with Ipilimumab plus Nivolumab in advanced Uveal Melanoma (CHOPIN).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 yrs
2. World Health Organization (WHO) Performance Status 0 or I
3. 50% or less histologically or cytologically confirmed unresectable metastatic uveal melanoma in the parenchyma of the liver
4. Hepatic metastases, confined to or predominantly in the liver
5. No prior systemic treatment (including chemotherapy, vaccine therapy, monoclonal Ab treatment, IL-2)
6. Local pre-treatment of uveal melanoma metastases is allowed (resection and/or thermal ablation), except for chemotherapy containing procedures (e.g. chemoembolization) and radio-embolization, and as long as patients have progressed with measurable disease according to RECIST 1.1
7. No concurrent systemic immunosuppressive medications ≥ 10mg/day prednisone or equivalent. Topical, inhaled, nasal and ophthalmic steroids, and adrenal replacement therapy are allowed.
8. Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥ 1.0x109/L, Platelets ≥ 100 x109/L, Hemoglobin ≥ 6.5 mmol/L, Creatinine ≤ 2x ULN, AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN, Total bilirubin ≤ 1.5 X ULN, INR and PTT in normal range, LDH < 2xULN
9. Women of child bearing potential (WOCBP) must agree to use a reliable form of contraceptive as described in paragraph 5.4.
10. Men must agree to the use of male contraception as described in paragraph 5.4.
11. Absence of additional severe and/or uncontrolled concurrent disease
12. No prior, or ongoing other malignancy, except adequately treated basal cell or squamous cell skin cancer, cervical cancer in situ or adequately treated other cancer with eradicative intent for which the patient has been continuously disease-free for > 2 years.
13. No aberrant vascular anatomy of the liver that precludes PHP

Exclusion Criteria:

1. Cerebral or meningeal metastasized uveal melanoma
2. Subjects with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy;
3. Prior immunotherapy (tumor vaccine, cytokine, or growth factor)
4. Known history of infection with Human Immunodeficiency Virus;
5. Active infection requiring therapy, positive serology for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA)
6. History of congestive heart failure, active cardiac conditions, including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia.
7. History or evidence of clinically significant pulmonary disease e.g. severe COPD that precludes the use of general anesthesia.
8. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study treatment hazardous or obscure the interpretation of toxicity determination or adverse events;
9. Latex allergy, and known hypersensitivity/allergy to ipilimumab, nivolumab, melphalan or heparin
10. Prior Whipple's Surgery
11. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids;
12. History of or current immunodeficiency disease, splenectomy or splenic irradiation; prior allogeneic stem cell transplantation;
13. Patients who are unable to be temporarily removed from chronic anti-coagulation therapy.
14. Patients with active bacterial infections with systemic manifestations (malaise, fever, leucocytosis) are not eligible until completion of appropriate therapy.
15. Use of other investigational drugs before study drug administration for systemic malignancy
16. Pregnancy or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity and safety of treatment | 36 weeks
  Dose limiting toxicities, maximum tolerated dose and recommended phase dose of the combination ipilimumab/nivolumab and PHP in patients with unresectable, histologically confirmed hepatic metastasis of uveal melanoma in phase Ib part.
Efficacy and safety | 1 year
  Description of PFS according to RECIST 1.1 at one year in the PHP group versus PHP + ipilimumab/nivolumab group in the phase II part.

SECONDARY OUTCOMES:
Response rate | 1 year
  Description of response rate and overall survival, overall clinical response, and duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W. Kapiteijn, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tong TML, van der Kooij MK, Speetjens FM, van Erkel AR, van der Meer RW, Lutjeboer J, van Persijn van Meerten EL, Martini CH, Zoethout RWM, Tijl FGJ, Blank CU, Burgmans MC, Kapiteijn E. Combining Hepatic Percutaneous Perfusion with Ipilimumab plus Nivolumab in advanced uveal melanoma (CHOPIN): study protocol for a phase Ib/randomized phase II trial. Trials. 2022 Feb 13;23(1):137. doi: 10.1186/s13063-022-06036-y. PMID 35152908